CLINICAL TRIAL: NCT02902263
Title: Inter-Hospital Transfer to a Vascular Neurology Unit After Telethrombolysis in France Comté
Brief Title: Inter-Hospital Transfer to a Vascular Neurology Unit After Telethrombolysis
Acronym: TRATT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2015/248
Record Dates: First submitted 2016-08-31; First posted 2016-09-15 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2016-09

CONDITIONS: Ischemic Stroke
Keywords: Telemedecine; Thrombolysis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Early thrombolysis is essential in treating ischemic strokes. The time window for thrombolysis is limited to 4,5 hours after symptoms onset.

In the French region of Franche Comté, in order to reduce the thrombolytic delay, a telemedicine network was developed between the neurovascular reference unit (NVU) localised in the University Hospital of Besançon and the peripheral hospital centres. Patients may then be transported to the NVU immediately after the thrombolysis initiation.

The aim of our study was to assess the relevance of a systematic medicalization of transfer to the NVU of patients with stroke who were telethrombolyzed before.

It was a retrospective, monocentric and observational study conducted over 24 months, in Franche-Comte (France).

DETAILED DESCRIPTION:
Stroke is a major health problem with increasing incidence. It represents the leading cause of disability and the third cause of death in France. There are two main types of stroke: ischemic (80%) or hemorrhagic (20%).

Early thrombolysis is essential in treating ischemic strokes. The time window for thrombolysis is limited to 4,5 hours after symptoms onset.

In the French region of Franche Comté, in order to reduce the thrombolytic delay, a telemedicine network was developed between the neurovascular reference unit (NVU) localised in the University Hospital of Besançon and the peripheral hospital centres. Patients may then be transported to the NVU immediately after the thrombolysis initiation.

The aim of our study was to assess the relevance of a systematic medicalization of transfer to the NVU of patients with stroke who were telethrombolyzed before.

It was a retrospective, monocentric and observational study conducted over 24 months, in Franche-Comte (France). Evaluation of neurological status was made with the Glasgow score (GCS) and National Institute of Health Stroke Score (NIHSS). The respiratory (SpO2; needs O2) and hemodynamic status (arterial blood pressure, heart rate) were assessed as well as the need for medical resuscitation at different times of the transport (thrombolysis, transfer, arrival at the Regional University Hospital Centre).

ELIGIBILITY:
Inclusion Criteria:

* Patient with ischaemic stroke
* Emergency department admission between 01/01/2012 and 12/31/2013
* Telemedicine stroke consult
* Thrombolysis therapy
* Patient transfered to NVU after thrombolysis initiation
* Transfer staffed by a qualified physician

Exclusion Criteria:

* Transfer non staffed by a qualified physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted in one emergency departments of four peripheral hospital centres in Franche Comté (Pontarlier, Vesoul, Gray and Dôle).
  Patients admitted for ischemic stroke, treated by thrombolysis and transferred to tue NVU
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Patient neurological status assessed by NIHSS score during transfer to NVU | one day
Patient neurological status assessed by Glasgow score during transfer to NVU | one day

SECONDARY OUTCOMES:
Patient respiratory status assessed by oxygen saturation | one day
Patient hemodynamic status assessed by systolic and diastolic pressure | one day

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nenert E, Pretalli JB, Bouamra B, Puyraveau M, Fehner L, Labourey JM, Desmettre T. Transfert interhospitalier vers une unité de neurologie vasculaire des accidents vasculaires cérébraux ischémiques téléthrombolysés : pertinence d'une médicalisation systématique ? Ann. Fr. Med. Urgence (2016).